CLINICAL TRIAL: NCT05894876
Title: A Study of the Genetic Determinants of Response to Growth Hormone Treatment in Children With Idiopathic Short Stature
Brief Title: A Study of the Genetic Basis of Response to Growth Hormone Treatment in Children With Idiopathic Short Stature
Status: Terminated | Type: Observational
Why Stopped: Due to recruitment challenges, the sponsor has decided to terminate the study prematurely.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-4978; U1111-1285-4921 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Short Stature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good responders: Participants on previous treatment with growth hormone will have one study visit for taking a non-invasive biological sample. Good responders are defined as participants with a change in height Standard Deviation Score (SDS) more than (>) 1.0, corresponding to >85th percentile.
  Interventions: Other: No treatment is given
- Poor responders: Participants on previous treatment with growth hormone will have one study visit for taking a non-invasive biological sample. Poor responders are defined as participants with a change in height SDS less than (<) 0.4, corresponding to <15th percentile.
  Interventions: Other: No treatment is given

INTERVENTIONS:
Other: No treatment is given — No treatment is provided to the participants as part of this study.

SUMMARY:
The study doctor will collect information from participants with Idiopathic Short Stature, who were treated with growth hormone for at least a year when they were children, before they reached puberty. The word "Idiopathic" refers to "unknown cause", and as such the study participants have/had short stature with no identifiable medical cause. The purpose of the study is to identify differences in the genetic characteristics of participants who responded well or poorly to growth hormone therapy. No medications or other treatments are provided to the participants by Novo Nordisk as part of this study. The study will last for up to 1 year. The participants will attend their usual doctor's appointments. If the participants are not usually visiting the clinic, they will need to do it only once as part of this study. If the participant agrees to take part in the study, they will be asked to read and sign the 'Agreement to take part form'.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent/parental consent and patient assent for minor children obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Patient has been diagnosed with Idiopathic Short Stature (ISS) and received at least 1 year of GH therapy.
* Patient was prepubertal at initiation of and throughout first year of GH therapy, as determined by the treating physician and patient medical records.
* Patient had no prior exposure to growth promoting therapy prior to initiation of GH therapy, including but not limited to growth hormone, IGF-I and ghrelin analogues.
* Age at initiation of GH therapy:

  * Boys: Age above or equal to 3 years and below 11.0 years.
  * Girls: Age above or equal to 3 years and below 10.0 years.
* Impaired height prior to initiation of GH therapy defined as at least 2 standard deviations below the mean height for chronological age and sex according to local growth reference charts. In the absence of local reference charts, the standards of Centres for Disease Control and Prevention should be used.
* GH deficiency has been excluded via GH stimulation test (cut point of 7 nanograms per milliliter [ng/ml]) or other clinical and biochemical criteria according to local clinical practice.
* Patient fits within one of the following response groups:

  * Change in Height Standard Deviation Score (SDS) after approximately the first year (+/- 2 months) of GH therapy greater than (>) 1.0.
  * Change in Height SDS after approximately the first year (+/- 2 months) of GH therapy less than (<) 0.4.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding, cooperation or informed consent.
* Receipt of any investigational medicinal product within 3 months before or during the first year of GH therapy that could influence response to GH therapy.
* Concomitant illness within 3 months before or during the first year of GH therapy that could (positively or negatively) influence the first year of GH therapy. Exception: Attention Deficit Hyperactive Disorder and its treatment can be included but should be recorded.
* Children with suspected or confirmed growth hormone deficiency according to local practice.
* Concomitant use of medication including gonadotropin-releasing hormone (GnRH) analogues, aromatase inhibitors, sex steroids, glucocorticoids or any other medication that can influence response to GH therapy. Exception: Attention Deficit Hyperactive Disorder and its treatment can be included but should be recorded.
* Any known or suspected clinically significant abnormality likely to affect growth or the ability to evaluate growth with standing height measurements, such as but not limited to:

  * Significant spinal abnormalities including but not limited to scoliosis, kyphosis and spina bifida variants.
  * Any other disorder that can cause short stature such as, but not limited to, psychiatric disorders, nutritional disorders, chronic systemic illness, chronic respiratory conditions (e.g. asthma), and chronic renal disease.
  * Turner Syndrome (including mosaicism).
  * Noonan Syndrome.
  * Born small for gestational age (defined as birth length below -2 SDS OR birth weight below -2 SDS OR both) (according to national standards).
  * Extreme prematurity, defined as gestational age less than 32 weeks.
  * Syndromic short stature defined by the presence of significant dysmorphic features and/OR major malformations, Laron syndrome, Prader-Willi syndrome, Russell-Silver syndrome.
  * Significant developmental delays, autism spectrum or intellectual deficit of any degree.
  * Skeletal dysplasia.
  * Magnetic resonance imaging (MRI) result confirming pituitary structural abnormalities.
  * Poor adherence to GH therapy or interruption of it for any time during the first year of therapy, as judged by the treating physician.

Ages: 3 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: Study population will consist of participants treated with GH for at least one year when they were prepubertal ISS children and had no prior exposure to growth promoting therapy prior to initiation of GH therapy, including but not limited to growth hormone, Insulin-like Growth Factor type 1 (IGF-1) and ghrelin analogues.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
The frequency of genetic variants that significantly differ between the two responder groups | One year after growth hormone therapy
  Measured as odds ratio.

SECONDARY OUTCOMES:
The enrichment of genetic variants per gene/pathway | One year after growth hormone therapy
  Measured as count.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (4):
- United States (2):
  - [Legal] Children's Hospital of Orange County on behalf of CHOC Children's Hospital of Orange County, Orange, California
  - Novo Nordisk Investigational Site, Columbia, Maryland
- University of Sao Paulo School of Medicine, São Pauloa, Brazil
- Assuta Ashdod Division of Pediatric Endocrinology and Diabetes, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com